CLINICAL TRIAL: NCT01648894
Title: Randomized Control Trial Comparing the Impact of a Lengthening of the Interval Between the Radiochemotherapy and Surgery (7 Weeks vs. 11 Weeks) on Complete Pathological Response in Rectal Cancer
Brief Title: Influence of Lengthening the Interval Between Radiochemotherapy and Surgery on Complete Pathological Response in Rectal Cancer
Acronym: GRECCAR6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 110125; AOM 11304 (Other: Assistance Publique)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; radiochemotherapy; complete pathological response
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 11 weeks (Experimental): The cancer surgery is practice 11 weeks after neoadjuvant radio-chemotherapy
  Interventions: Procedure: Surgery after 11 weeks of delay after chemoradiotherapy.
- 7 weeks (Other): The cancer surgery is practice 7 weeks after neoadjuvant radio-chemotherapy
  Interventions: Procedure: Surgery after 7 weeks of delay after chemoradiotherapy

INTERVENTIONS:
Procedure: Surgery after 11 weeks of delay after chemoradiotherapy. — Surgery consists carcinological resection of the rectal cancer with total excision of the mesorectum after 11 weeks of delay after the end of chemoradiotherapy.
  Arms: 11 weeks
Procedure: Surgery after 7 weeks of delay after chemoradiotherapy — Surgery consists carcinological resection of the rectal cancer with total excision of the mesorectum after 7 weeks of delay after the end of chemoradiotherapy
  Arms: 7 weeks

SUMMARY:
At the end of the neoadjuvant radiochemotherapy, patients are seen by their surgeon to planify the surgery. During this visit, the study will be explained them and their consent obtained. They will then be randomized between the two groups 7 weeks vs. 11 weeks. Patients were reviewed 15 days before surgery and at 1 and 3 months after surgery. Participation in this study does not change treatment, investigations and consultations usually necessary for management of rectal cancer. The objective is to improve the pathological complete response rate of the rectal cancer.

DETAILED DESCRIPTION:
D0: Visit of inclusion and randomization After the end of chemoradiotherapy, the patient is seen in consultation by her / him a surgeon who propose him to participate in the study. At the end of the visit if the patient agrees to participate in it, the investigator at each center will conduct the collection of written consent to the inclusion of the patient. Inclusion will be recorded in the electronic Case Report Form (e-CRF) by the investigator at each center. Randomization (7 or 11 weeks of delay) is performed by the surgeon via the software module CleanWeb randomization.

M1- 1.5 or M2.5 depending of the group randomisation A consultation with the surgeon is held within 15 days (+/- 5 days) of intervention to check the clinical response (tumor regression in rectal tumor distance from the dentate line) and planify surgery. During this visit, the surgeon noted in the e-CRF, clinical findings of the lesion and the results of further investigations.

Not specific exam is requested in the study.

M2 or M3

Surgical procedure:

The anesthesia consultation is planned before the surgery according to the habits of service. Participation in the study does not alter the anesthetic procedures.The patient is admitted the day before surgery in the surgical ward.

During surgery, the operating data are provided on the e-CRF (digital rectal examination under general anesthesia, type of surgery (anterior resection or abdominal-perineal resection), operative time, intraoperative bleeding, macroscopic appearance of the mesorectum, distance from the distal limit of resection). The postoperative complications are noted by the surgeon in the e-CRF during hospitalization (about 10-15 days), and data reporting pathological (Annex 2).

Pathological examination of the specimen of proctectomy is performed according to recommendations for clinical practice using the standard form (Annex 2). The tumor response is evaluated by inclusion of all residual tumor and the response to chemoradiotherapy is graded with the scale of Rödel (Annex 5). A double reading of slides will be made for each patient by two independent pathologists blinded to the randomization group of the patient.

M2 - M5 or M3 - M6 :

Postoperative follow-up :

Following the intervention, no specific consultation is necessary. At follow-up consultations (1 month, 3 months) the surgeon evaluate the postoperative course, planify the stoma closure, noted the potential adverse events and results of morphological examinations (computed tomography, ultrasound, endoscopy) and biological (markers) eventually prescribed.

M6 - M60 :

Cancer surveillance :

Regular follow-up every 3-4 months fo the first two years and every 6 months for the last remaining 3 years (clinical examination, CT-scan and biological marker (CEA))

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years, no age limit higher
* Performance status evaluated by the Eastern CooperativeOncology Group (ECOG) score: 0-1,
* Patients with cancer of the middle or lower rectum (lesion located within 10 cm from the dentate line or 12 cm from the anal margin) proved by pathology,
* T3-T4N0, TxN+ on ultrasound-endoscopy and MRI, without secondary localization (M0) on the thoracoabdominal (or chest radiography and abdominal ultrasound)
* Patient who received a protocol between 45-51 Gy of radiotherapy and chemotherapy based on 5-fluorouracil for an average duration of 5 weeks for the management of rectal cancer,
* Curative surgical treatment planned following radiochemotherapy with total mesorectal excision,
* Free and informed consent signed by the patient,
* Patient affiliated to a social security scheme or beneficiary of such plan(except AME)
* Patient able, according to the investigator, to comply with the requirements of the study.

The cessation of chemotherapy during radiotherapy does not exclude the patient from the study.

Exclusion Criteria:

* Patient with metastasis,
* T1 or T2N0 tumor classified by echo-endoscopy and MRI,
* rectal tumor with lower pole is more than 12 cm from the anal margin or 10 cm from the dentate line,
* Patient did not complete the full protocol of radiotherapy,
* History of tumors (other than basal cell carcinoma and / or carcinoma in situ of the cervix) old less than 10 years
* A patient with impaired or incompetent investigator by not allowing him a good understanding of the requirements of the study,
* Person under guardianship, persons under guardianship, persons deprived of their liberty by judicial or administrative body, adult subject to legal protection or unable to consent,
* Patient did not complete the full protocole of chemotherapy,
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2012-10-25 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Percentage of pathological complete response after pathological examination of surgical specimen defined by the absence of persistent tumor cell invasion and lymph node (ypT0N0) in group 7 weeks versus 11 weeks in the group | 6 month

SECONDARY OUTCOMES:
Rates of clinical response to radio-chemotherapy before surgery, comparison between the two groups (7 versus 11 weeks) | 6 month
Rate of tumor regression, comparison between the two groups (7 versus 11 weeks) | 6 month
Rates of operative mortality and morbidity at 90 days, comparison between the two groups (7 versus 11 weeks) | 6 month
Quality of mesorectum resection, comparison between the two groups (7 versus 11 weeks) | 6 month
Rate of sphincter preservation, comparison between the two groups (7 versus 11 weeks) | 6 month
Local and distant recurrence rates, comparison between the two groups (7 versus 11 weeks) | 5 years
Overall survival and disease-free survival rates, comparison between the two groups (7 versus 11 weeks) | 5 years
Functional results (LARS score) | 24 months and 36 months
  LARS questionnaire (Low Anterior Resection Syndrome questionnaire) completed at 24 months and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Lefèvre, MD, Principal Investigator — Assistance Publique
Locations (1):
- Saint-Antoine Hospital - AP-HP, Department of general and digestive surgery, Paris, France

REFERENCES:
- [Derived] Lefevre JH, Mineur L, Kotti S, Rullier E, Rouanet P, de Chaisemartin C, Meunier B, Mehrdad J, Cotte E, Desrame J, Karoui M, Benoist S, Kirzin S, Berger A, Panis Y, Piessen G, Saudemont A, Prudhomme M, Peschaud F, Dubois A, Loriau J, Tuech JJ, Meurette G, Lupinacci R, Goasgen N, Parc Y, Simon T, Tiret E. Effect of Interval (7 or 11 weeks) Between Neoadjuvant Radiochemotherapy and Surgery on Complete Pathologic Response in Rectal Cancer: A Multicenter, Randomized, Controlled Trial (GRECCAR-6). J Clin Oncol. 2016 Nov 1;34(31):3773-3780. doi: 10.1200/JCO.2016.67.6049. PMID 27432930
- [Derived] Lefevre JH, Rousseau A, Svrcek M, Parc Y, Simon T, Tiret E; French Research Group of Rectal Cancer Surgery (GRECCAR). A multicentric randomized controlled trial on the impact of lengthening the interval between neoadjuvant radiochemotherapy and surgery on complete pathological response in rectal cancer (GRECCAR-6 trial): rationale and design. BMC Cancer. 2013 Sep 12;13:417. doi: 10.1186/1471-2407-13-417. PMID 24028546
- See also: Effect of Interval (7 or 11 weeks) Between Neoadjuvant Radiochemotherapy and Surgery on Complete Pathologic Response in Rectal Cancer: A Multicenter, Randomized, Controlled Trial (GRECCAR-6) — https://www.ncbi.nlm.nih.gov/pubmed/27432930